CLINICAL TRIAL: NCT06186934
Title: Post Marketing Surveillance Study to Observe Safety and Effectiveness of NEPHOXIL ® in S. Korea Patients
Status: Recruiting | Type: Observational
Sponsor: Kyowa Kirin Korea Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Kyowa Kirin Co., Ltd. (Industry)
Other Study IDs: Nephoxil PMS
Record Dates: First submitted 2023-12-17; First posted 2024-01-02 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Hyperphosphatemia
MeSH Terms: conditions — Hyperphosphatemia | interventions — Population Groups

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Weeks
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: the standard-dose group (4 g/day) — Patients with chronic kidney disease undergoing hemodialysis and controlling hyperphosphatemia

SUMMARY:
The objective of this post-marketing surveillance (PMS) study is to assess the safety and effectiveness of Nephoxil capsule 500 mg (Ferric Citrate 500 mg, equivalent to 105 mg Ferric Iron) in routine clinical settings

ELIGIBILITY:
Inclusion Criteria:

1. Adults 19 years of age or older
2. CKD patients undergoing hemodialysis to whom Nephoxil capsule administration is deemed necessary for improvement of hyperphosphatemia as per the determination of the investigator
3. Patients who received Nephoxil capsule for the first time according to the national approval after conclusion of the contract with the study institution
4. Those (or his / her legal guardian) who have agreed in writing to participate in the survey

Exclusion Criteria:

1. Patients with contraindications to receive Nephoxil

   * Patients with hypersensitivity to the active substance or to any of the excipients
   * Patients with hypophosphatemia
   * Patients with abnormal iron metabolism or symptoms of excessive iron (e.g. hemochromatosis)
2. Patients who intend to use this drug for non-approved indications
3. Patients who participated in pre-market clinical trials with Nephoxil
4. Patients who took this drug before the starting day of this survey

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with chronic kidney disease undergoing hemodialysis and controlling hyperphosphatemia
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2023-12-21 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Serum phosphorus levels | 8 weeks
  Effectiveness evaluation is performed based on Serum phosphorus levels (mg/dL) before and after Nephoxil administration. We collect the most recent measurements prior to the initial administration, and measurements after at least four and eight weeks of administration of Nephoxil

CONTACTS AND LOCATIONS:
Locations (1):
- Jesus Hospital, Jeonju, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
Undecided